CLINICAL TRIAL: NCT06636448
Title: The Effect of Body Mass Index on Patient Outcomes During Low-flow Anaesthesia for Major Gynaecological Cancer Surgery: a Prospective Observational Study
Brief Title: The Relationship Between Body Mass Index and Patient Outcomes in Low Flow Anaesthesia
Status: Completed | Type: Observational
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Duygu Akyol, Principal investigator, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Other Study IDs: 2024-04
Record Dates: First submitted 2024-09-27; First posted 2024-10-10 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2024-09

CONDITIONS: Major Gynecological Cancer Surgery; Low Flow Anesthesia
Keywords: major gynecological cancer surgery; low flow aneshesia; cerebral oxygenation; hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- obese patients undergoing low-flow anaesthesia: Low-flow anaesthesia was performed in patients with a body mass index between 30-40
  Interventions: Procedure: the effect of body mass index during low-flow anesthesia

INTERVENTIONS:
Procedure: the effect of body mass index during low-flow anesthesia — The investigator planned to evaluate the effect of body mass index on patient outcomes during low-flow anesthesia in patients undergoing gynecologic cancer surgery.

SUMMARY:
This study was designed as a prospective observational study.

DETAILED DESCRIPTION:
In this study, it was planned to evaluate the effect of body mass index on patient outcomes during low flow anaesthesia in patients undergoing gynaecological cancer surgery on the specified dates. ASA II and III patients over 18 years of age were included in the study. Low flow anaesthesia is routinely applied in open gynaecological cancer surgeries in our clinic. The relationship between body mass index and intraoperative haemodynamic and mechanical ventilator values and postoperative patient outcomes will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASA II-III
* >18 years
* Patients undergoing major open surgery for endometrium, cervix or ovarian ca in gynaecological oncology clinic

Exclusion Criteria:

* Patients who refused to participate in the study
* Cerebrovascular disease
* Those with severe pulmonary disease
* Those with serious cardiovascular disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: A total of 40 patients were planned for this study
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
postoperative hospital stay | up to 10 days postoperative
  The primary aim of this study was to evaluate the duration of postoperative hospital stay

OTHER OUTCOMES:
Intraoperative cerebral oxygenation | intraoperative process
  Our other aim was to evaluate right and left hemisphere cerebral oxygenation at certain time periods.

CONTACTS AND LOCATIONS:
Locations (1):
- Duygu, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mychaskiw G 2nd. Low and minimal flow anesthesia: Angels dancing on the point of a needle. J Anaesthesiol Clin Pharmacol. 2012 Oct;28(4):423-5. doi: 10.4103/0970-9185.101883. No abstract available. PMID 23225917
- [Background] Oterkus M, Donmez I, Nadir AH, Rencuzogullari I, Karabag Y, Binnetoglu K. The effect of low flow anesthesia on hemodynamic and peripheral oxygenation parameters in obesity surgery. Saudi Med J. 2021 Mar;42(3):264-269. doi: 10.15537/smj.2021.42.3.20200575. PMID 33632904
- [Background] Akbas S, Ozkan AS. Comparison of effects of low-flow and normal-flow anesthesia on cerebral oxygenation and bispectral index in morbidly obese patients undergoing laparoscopic sleeve gastrectomy: a prospective, randomized clinical trial. Wideochir Inne Tech Maloinwazyjne. 2019 Jan;14(1):19-26. doi: 10.5114/wiitm.2018.77265. Epub 2018 Jul 24. PMID 30766625